CLINICAL TRIAL: NCT04338074
Title: Exploratory Studies of the Effect of Tranexamic Acid Treatment on the Progression of COVID19 in Outpatients
Brief Title: TXA and Corona Virus 2019 (COVID19) in Outpatients
Acronym: TCOutpatient
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Timothy Ness, MD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TXACOVID1
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind comparison
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy prepares 5 day packs of medications that are coded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid Treatment (Experimental)
  Interventions: Drug: Tranexamic acid tablets
- Placebo Treatment (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Tranexamic acid tablets — Oral dosing of 1300 mg p.o. three times per day x 5 days versus identical placebos
  Arms: Tranexamic Acid Treatment
Drug: Placebo oral tablet — 2 tablets p.o. three times per day x 5 days
  Arms: Placebo Treatment

SUMMARY:
A controlled trial of the drug tranexamic acid (TXA) in outpatients who were recently diagnosed with COVID-19. It is hypothesized that TXA will reduce the infectivity and virulence of the virus.

DETAILED DESCRIPTION:
A recent report in Physiological Reviews proposed that the endogenous protease plasmin acts on the COVID19 virus by cleaving a newly inserted furin site in the S protein portion of the virus resulting in increased infectivity and virulence. Patients with hypertension, diabetes, coronary artery disease, cerebrovascular illness, lung disease and kidney dysfunction commonly have elevated levels of plasmin/plasminogen and it was proposed that this may be the mechanism for poorer outcomes in patients with these co-morbidities. A logical treatment that might blunt this process would be the inhibition of the conversion of plasminogen to plasmin. There is an inexpensive, commonly used drug, tranexamic acid, (TXA), which suppresses this conversion and could be re-purposed for the treatment of COVID19.

TXA is a synthetic analog of the amino acid lysine which reversibly binds four to five lysine receptor sites on plasminogen. This reduces conversion of plasminogen to plasmin, and is normally used to prevent fibrin degradation. TXA is FDA approved for treatment of heavy menstrual bleeding (typical dose 1300 mg p.o. three times per day x 5 days) and off-label use for many other indications. TXA is used perioperatively as a standard-of-care at the University of Alabama at Birmingham (UAB) for orthopedic and cardiac bypass surgeries. At our institution, it is commonly employed in hemorrhaging trauma patients and currently is being studied for perioperative use in Cesarean section surgeries. It has also been utilized for spinal surgery, neurosurgery, orthognathic surgeries and even long term for the treatment of cosmetic dermatological disorders with a long track record of safety. Given the potential benefit and limited toxicity of TXA it would appear warranted to perform a rapid randomized, double-blind placebo controlled exploratory trial at UAB in the treatment of the early phases of COVID19 to determine whether it reduces infectivity and virulence of the COVID19 virus as hypothesized. Involvement of each patient is only for 7 days before primary endpoints.

An exploratory, randomized, placebo-controlled, double-blind Phase 2 clinical trial in which study patients have just been diagnosed with COVID19 as an outpatient. The overall goal of this exploratory study is to assess both safety and efficacy of 5 days of TXA versus placebo in the COVID19 population. All patients would also receive apixaban 5 mg p.o. BID. The primary endpoint for the study would be a need for hospitalization. Contact would consist of daily phone contact. Care for COVID19 would otherwise be standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID-19 test
* Outpatient
* Age >/= 19 y.o.

Exclusion Criteria:

* Allergic reaction to tranexamic acid
* History of hypercoagulation disorders (deep venous thrombosis, pulmonary thromboembolism)
* Ongoing anticoagulation
* History of GI bleeding
* History of Seizures
* Cardiac or other vascular stents
* History of severe renal disease
* History of intracranial hemorrhage

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Ness, MD PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid Treatment | Placebo Treatment
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 38 [32 to 45] | 37 [34 to 40] | 38 [32 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Hospitalization
Description: Participant admission to hospital for COVID-19 treatment
Time Frame: Randomization to 7 days after randomization
Population: Categorical data - admitted to hospital or not
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Treatment | Placebo Treatment
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days after onset of treatment
Description: There were no adverse events related to drug treatment in this truncated trial
Arm/Group | Tranexamic Acid Treatment | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT04338074/Prot_SAP_003.pdf